CLINICAL TRIAL: NCT01108276
Title: A Prospective, Randomized, Controlled Study Comparing the Efficacy of the ConvaTec Engenex® Negative Pressure Wound Therapy (NPWT) Device to Moist Wound Therapy (MWT) in the Treatment of Diabetic Foot Wounds
Brief Title: Comparing the Efficacy of the ConvaTec Engenex® Negative Pressure Wound Therapy Device to Moist Wound Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started and therefore terminated.
Sponsor: Georgetown University (Other)
Collaborators: ConvaTec Inc. (Industry)
Responsible Party: Principal Investigator, John Steinberg, DPM, Associate Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-071
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes; Foot Wound
MeSH Terms: conditions — Diabetes Mellitus; Foot Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Convatec engenex negative pressure wound therapy — ConvaTec Engenex® is a negative pressure wound therapy that stimulates wound healing and promotes granulation tissue formation, removal of wound exudate and infectious materials by the application of negative pressure to wounds. It utilizes Bio-Dome™ Dressing technology to effectively control infection, drainage and odor while promoting granulation and wound healing at 75mmHg pressure.
  Other Names: Convatec engenex

SUMMARY:
This is an investigator-initiated prospective, randomized, controlled study. Hypothesis/Objective: The study will evaluate the rates of wound healing among patients with lower extremity diabetic wounds comparing two groups of patients. Group 1, the control group, will be treated with the standard of care treatment of moist wound therapy. Group 2 will be treated with ConvaTec Engenex® NPWT. Both groups will be treated in the inpatient and outpatient setting. It is expected that the NPWT device will be an effective therapy that expedites time to closure and demonstrates a significant decrease in the size and depth of the wound over the course of the 12 week therapy as compared to the standard of care.

DETAILED DESCRIPTION:
After determining if you meet the criteria to be included in the study, your wound will be debrided (cleansed of any dead tissue or infection). You will then be randomly placed into one of two treatment groups. Group 1 will be the control group and a moist wound therapy will be applied to the wound. Either you or home nursing will then change the dressing twice a week. Group 2 will have a negative pressure wound therapy (NPWT) dressing applied. The NPWT dressing will be changed twice a week by home nursing. You will return to clinic every 2 weeks for a total of 12 weeks for observation and assessment of the diabetic foot ulcer. If wound healing occurs prior to 12 weeks, a final assessment visit will be done and the status of the healed ulcer will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older
2. Subjects with chronic lower extremity diabetic wounds, with or without a previous history of partial foot amputation.
3. Subject has Diabetes Mellitus (type 1 or type 2)
4. University of Texas Classification 1A-3A or 1B-3B
5. Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study.

Exclusion Criteria:

1. Subjects < 18 years of age
2. Subject is non-diabetic
3. Subjects who present with wounds of etiology other than diabetes
4. Subject demonstrates increased signs of clinical infection
5. Has active malignant disease of any kind. A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
6. University of Texas Classification 1C-3C
7. Subjects participating in any other trials in regards to the diabetic foot ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Overall decrease in wound size | 12 weeks
  Overall decrease in wound size, summary statistics will be performed comparing both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: John Steinberg, DPM, Principal Investigator — Georgetown University Hospital